CLINICAL TRIAL: NCT06421064
Title: Clinical Profile and Surgical Treatment Outcome of Perforated Peptic Ulcer Disease in Public Hospitals of Eastern Ethiopia: a Prospective Multicenter Study.
Brief Title: Clinical Profile and Outcome of Perforated PUD
Acronym: PUD
Status: Completed | Type: Observational
Sponsor: Badhaasaa (Other)
Responsible Party: Sponsor-Investigator, Badhaasaa, Assistant professor, Haramaya Unversity
Organization: Haramaya Unversity (Other)
Other Study IDs: HURG-2020
Record Dates: First submitted 2024-05-10; First posted 2024-05-20 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Diseases or Conditions
MeSH Terms: conditions — Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Perforation repair — All patients were operated with slight difference but all had perforation repaired.

SUMMARY:
Perforated peptic ulcer disease (PPUD) is series illness that need emergency intervention. Its overall clinical profile and treatment outcome was also not well studied in developing countries. Therefore the study was aimed to see the outcome of surgical intervention and associated factors.

The study was a retrospective observational study conducted using the medical records of patients operated on for perforated peptic ulcer disease at a multicenter, in eastern Ethiopia.

DETAILED DESCRIPTION:
This study was designed to investigate the clinical characteristics and treatment outcomes among adult patients presented to the study areas. Three teaching Hospitals and one Regional Hospital were chosen and data collection was effected for two years. One hundred seventy patients participated in this observational study.

ELIGIBILITY:
Inclusion Criteria:

* All adults with a diagnosis of perforated PUD managed at HU until discharged

Exclusion Criteria:

* Patients who were referred to other institutions before official discharge, Incomplete Medical record

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All surgical emergency admissions.
Sampling Method: Non-Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Survival outcome of perforated PUD | 2 years
  This is a dichotomous variable, either survived or deceased.

CONTACTS AND LOCATIONS:
Locations (1):
- Haramaya University, Harar, Ethiopia

IPD SHARING:
Plan to Share IPD: No
Owned by the university